CLINICAL TRIAL: NCT00889538
Title: Double-Blind, Placebo-Controlled, Crossover Study of Glutathione, Vitamin C and Cysteine in Children With Autism and Severe Behavior Problems
Brief Title: Study of Glutathione, Vitamin C and Cysteine in Children With Autism and Severe Behavior Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Cumberland Pharmaceuticals (Industry); Norton Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Glutathione-KCPCRU-01
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Autism; Severe Behavior Disorder
Keywords: Autism; Severe Behavior Disorder; Glutathione; Antioxidants
MeSH Terms: conditions — Autistic Disorder; Mental Disorders | interventions — Glutathione; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Randomized to placebo or treatment (glutathione or glutathione/vit C/NAC)
  Interventions: Drug: placebo
- Glutathione (Active Comparator): Randomized to placebo or treatment (glutathione or glutathione/vit C/NAC)
  Interventions: Drug: glutathione
- Glutathione, Vit C and NAC (Active Comparator): Randomized to placebo or treatment (glutathione or glutathione/vit C/NAC)
  Interventions: Drug: glutathione, vit C and NAC

INTERVENTIONS:
Drug: placebo — 50 mL of 1/2 normal saline IV
  Arms: Placebo
Drug: glutathione — glutathione 600 mg IV
  Arms: Glutathione
Drug: glutathione, vit C and NAC — Glutathione 600 mg IV Vitamin C 2000 mg IV N-acetylcysteine 20 mg/kg IV (max dose = 600 mg) Mix above three in 1/2 NS for a total volume of 50 mL
  Other Names: NAC
  Arms: Glutathione, Vit C and NAC

SUMMARY:
This is a double-blind, placebo-controlled crossover study to evaluate the safety and efficacy of glutathione alone or glutathione, vitamin C and NAC treatment in children with autism who also have severe behavior problems. The investigators hypothesis is that children with autism will show improvement in both learning capabilities and behavior with either glutathione, or glutathione, vitamin C and NAC therapy.

DETAILED DESCRIPTION:
This is a prospective, single center, double-blind, randomized pilot study in children and adolescents with autism and severe behavior disorders. All subjects will undergo initial screening procedures to determine eligibility. They will then be randomized to either 8 weeks of placebo or 8 weeks of glutathione or glutathione, vitamin C and N-acetylcysteine. They will receive intravenous treatment weekly and will have ongoing behavioral studies during this period. Following 8 weeks of therapy, they will have a week without treatment then will cross-over to the alternate therapy for weekly intravenous infusions and behavioral testing. In addition to baseline hematology and chemistries, baseline oxidized and reduced glutathione will be measured. These parameters will be repeated at the end of each 8 week course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 to 16 years, inclusive
* Diagnosed with autism using the ADI-R (Autism Diagnostic Interview-Revised)
* ABC Irritability/Agitation subscale score (Aberrant Behavior Checklist Subscale) ≥ 18
* CGI-S score (Clinical Global Impression-Severity Scale) ≥ 4
* Must be drug naïve or on a stable dose of medication(s) and educational/behavioral interventions for one month prior to participation
* Parent/legal guardian must provide written consent and required research authorization (i.e. HIPAA) prior to the performance of any study procedures.

Exclusion Criteria:

* Presence of another disorder on the autism spectrum including PDD-NOS (Pervasive Developmental Disorder Not Otherwise Specified), Asperger's, and Rett's Syndrome
* Patient with a known cause of autism such as Fragile X
* Evidence of significant renal dysfunction (e.g. GFR estimated by the Schwartz formula < 50 mL/min or serum creatinine > 2.5 X upper limit of normal for age)
* Evidence of significant hepatic dysfunction (serum transaminases > 2.5 X the upper limit of normal)
* Known hypersensitivity to glutathione, vitamin C or NAC
* Pregnant or lactating female
* Inability of subject and parent to be able to comply with requirements for study visits and procedures
* Presence of major mental illness
* History of antioxidant supplementation.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Improvement in both developmental skills and behavior with either glutathione or glutathione, Vitamin C and N-acetylcysteine therapy as compared to placebo therapy. Subjects will also be monitored using clinical and laboratory safety parameters. | 4 months
  Improvement in both developmental skills and behavior measured using validated scales in subjects receiving either glutathione, glutathione/Vitamin C/N-acetylcysteine or placebo measured at baseline, 9 weeks and at the end of study in a double-blind cross-over design.

SECONDARY OUTCOMES:
Response to glutathione (changes in behavior) will correlate with the glutathione level (GSH) and GSH:GSSG ratio | Baseline
Response to glutathione (changes in behavior) will correlate with the glutathione level (GSH) and GSH:GSSG ratio | 9 weeks
Response to glutathione (changes in behavior) will correlate with the glutathione level (GSH) and GSH:GSSG ratio | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patricia G. Williams, MD, Principal Investigator — University of Louisville; Janice E. Sullivan, M.D., Study Director — University of Louisville
Locations (1):
- KCPCRU, Louisville, Kentucky, United States